CLINICAL TRIAL: NCT03897153
Title: Evaluation of the SONAS® Ultrasound Device for the Assessment of Bilateral Cerebral Perfusion in Subjects With Acute Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Burl Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SONAS2018
Record Dates: First submitted 2019-03-28; First posted 2019-04-01 (Actual); Last update posted 2019-04-01 (Actual); Status verified 2019-03

CONDITIONS: Stroke, Acute
Keywords: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental:Diagnostic (Experimental): Diagnostic Test: SONAS® Ultrasound Device
  Interventions: Device: SONAS® Ultrasound Device

INTERVENTIONS:
Device: SONAS® Ultrasound Device — The SONAS® Ultrasound Device is intended for non-invasive transcranial ultrasound and used with a commercially approved contrast agent (e.g., Lumason®/SonoVue®).

SUMMARY:
The purpose of this clinical investigation is to determine the safety and feasibility of detecting acoustic signals related to blood supply in subjects with acute large vessel occlusion (LVO) stroke by using the SONAS® device.

DETAILED DESCRIPTION:
This clinical investigation will assess the performance of the SONAS® device in subjects with acute stroke admitted to the emergency department or stroke unit within 24 hours of symptoms onset and confirmed occlusion of either the proximal middle, distal M1-segment cerebral arteries, or distal internal carotid arteries (including carotid-T occlusion) by cerebral magnetic resonance imaging (cMRI) or cerebral imaging computed tomography (cCT), including perfusion weighted (pw) imaging sequences, will be considered for the investigation.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained
2. Male or female subject ≥18 years
3. Clinical diagnosis of acute stroke (NIHSS score: ≥10)
4. Time of stroke symptoms onset: ≤24 hours
5. Confirmed occlusion of either the proximal middle cerebral artery (occlusion of the proximal, middle or distal M1-segment) or the distal internal carotid artery (including carotid-T occlusion) by cMRI or cCT (including perfusion weighted imaging sequences)
6. Women of childbearing potential must have a negative urine or serum beta human chorionic gonadotropin result, obtained within 24 hours before administration of SonoVue®
7. Women of non-childbearing potential can be included in the clinical investigation, if confirmed by fulfilling at least 1 of the following criteria:

   * Postmenopausal (age-related amenorrhea for ≥12 consecutive months)
   * Documentation (based on medical records, medical examination, or medical history interview) of irreversible surgical sterilization by bilateral oophorectomy, bilateral salpingectomy, or hysterectomy

Exclusion Criteria:

1. Subjects with known contraindications to the use of SonoVue®:

   * Subjects known to have right-to-left shunts, severe pulmonary hypertension (pulmonary artery pressure >90 mmHg), uncontrolled systemic hypertension, and subjects with acute respiratory distress syndrome
   * SonoVue® must not be used in combination with dobutamine in subjects with conditions suggesting cardiovascular instability where dobutamine is contraindicated
   * Known hypersensitivity to any of the following substances:

     * Sulphur hexafluoride
     * Macrogol 4000
     * Distearoylphosphatidylcholine
     * Dipalmitoylphosphatidylglycerol sodium
     * Palmitic acid
2. Pregnant women
3. Subjects with severe cardiac or pulmonary disease as defined by the treating physician
4. Subjects with acute endocarditis and/or artificial heart valve
5. Subjects with acute systemic inflammation and/or sepsis
6. Subjects with hyperactive coagulation states and/or a recent thromboembolism
7. Subjects with end stage renal or hepatic disease
8. Subjects with known metal skull implants in the anatomical area of the temporal/parietal bones, or with anatomical formation of the head or ear that may interfere with proper headset placement, or with significant observable asymmetry in head formation
9. Subjects with known implanted deep brain stimulation devices
10. Subjects with known or suspected fracture(s) of the temporal/parietal skull bones, or with open skin injuries in the anatomical area of the temporal/parietal lobes
11. Subjects with known significant blood loss prior to or during the test procedure, SONAS® should not be used unless the blood pressure of the subject is verified to be stabilized
12. Subjects with axial (coronal) skull diameters of <12 cm or >18 cm
13. Subjects participating in another clinical investigation with an investigational drug or device within 3 months of enrollment or planned participation at any time during this clinical investigation
14. Previous participation in this clinical investigation
15. Employees of the clinical investigation site or the sponsor directly involved with the conduct of the clinical investigation, or immediate family members of any such individuals
16. Subjects committed to an institution by an order issued either by the courts or by an authority

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-02-12 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-10 (Estimated)

PRIMARY OUTCOMES:
Assessment of Brain Perfusion | 24 hours
  Measurement of the kinetic parameter time to peak (TTP) in the right and left-brain hemisphere during the SONAS® test
Comparison | 7 days
  Comparison between SONAS® versus cMRI or cCT generated intra-individual differences in the parameter TTP in the right and left-brain hemisphere
Assessment of Adverse Events | 72 hours
  Frequency, severity, relationship (to device, contrast agent, or procedure), and outcome of AEs Frequency, severity, relationship (to device, contrast agent, or procedure), and outcome of AEs Frequency, severity, relationship (to device, contrast agent, or procedure), and outcome of AEs

CONTACTS AND LOCATIONS:
Locations (2):
- Universitätsklinik für Neurologie / Medizinische Universität Wien, Vienna, Austria
- Universitätsklinik für Neurologie / Universitätsklinikum Regensburg, Regensburg, Germany

IPD SHARING:
Plan to Share IPD: No